CLINICAL TRIAL: NCT06824051
Title: A Phase 1, Double-blind, Two-arm, Mechanism of Action Study to Investigate the Effect of Orforglipron on Body Composition in Adult Participants With Obesity or Overweight, Without Diabetes
Brief Title: A Study of Orforglipron (LY3502970) in Adult Participants With Obesity or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27352; J2A-MC-GZPQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-01-27; First posted 2025-02-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
Keywords: Visceral adipose tissue; Energy intake
MeSH Terms: conditions — Obesity; Overweight | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orforglipron (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to see how orforglipron affects the amount of body fat compared with placebo in participants with obesity or overweight. Participation in the study will last approximately 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index (BMI)

  * ≥30.0 kilograms per square meter (kg/m2), or
  * ≥27.0 kg/m2 with comorbidities

Exclusion Criteria:

* Have type 1 diabetes, type 2 diabetes, or any other types of diabetes, history of ketoacidosis, or hyperosmolar state/coma
* Have an unstable body weight within 90 days prior to screening
* Have acute or chronic hepatitis
* Are taking other medications or alternative remedies to manage weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Visceral Adipose Tissue (VAT) | Baseline, Week 36

SECONDARY OUTCOMES:
Percent Change from Baseline in Energy Intake | Baseline, Week 36
Percent Change from Baseline in Appetite | Baseline, Week 36
Percent Change from Baseline in Body Weight | Baseline, Week 36
Percent Change from Baseline in Fasting Total Cholesterol | Baseline, Week 36
Percent Change from Baseline in High-Sensitivity C-Reactive Protein (hs-CRP) | Baseline, Week 36
Change from Baseline in International Physical Activity Questionnaire-Long Form (IPAQ-L) Scores | Baseline, Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 : Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Axis, Dilworth, Minnesota
  - Ohio Clinical Trials, Columbus, Ohio
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Orforglipron (LY3502970) in Adult Participants with Obesity or Overweight — https://trials.lilly.com/en-US/trial/575755